CLINICAL TRIAL: NCT07120529
Title: Minimally Invasive Surgery Versus Open Radical Hysterectomy in Presumably Early Stage Cervical Cancer: a Retrospective Multicenter Non-inferiority Study Comparing Overall and Progression-free Survival.
Acronym: MOOSE
Status: Recruiting | Type: Observational
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Krzysztof Nowosielski, Prof., Medical University of Silesia
Other Study IDs: BNW/NWN/0052/KB/59/25
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cervical Cancer; Hysterectomy
Keywords: cervical cancer; radical laparoscopic hysterectomy; radical abdominal hysterectomy; protective maneuver; LACC study
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RLH: Radical laparoscopic hysterectomy
  Interventions: Other: CT scan; Procedure: Ultrasound scan (Transvaginal or Transabdominal); Procedure: Gynecological examination
- RAL: Radical open hysterectomy
  Interventions: Other: CT scan; Procedure: Ultrasound scan (Transvaginal or Transabdominal); Procedure: Gynecological examination

INTERVENTIONS:
Other: CT scan — CT chest, abdominal, pelvis during follow-up
Procedure: Ultrasound scan (Transvaginal or Transabdominal) — Transvaginal and transabdominal ultrasound scan during follow-up
Procedure: Gynecological examination — Gynecological standard examination during follow-up

SUMMARY:
The goal of this retrospective observational study with prospective follow-up is to compare the safety and treatment outcomes of radical laparoscopic hysterectomy (removal of the uterus with cervix) versus abdominal (open) hysterectomy performed after the publication of the LACC trial in women with early-stage cervical cancer.

Eligible participants will include adult, legally competent women diagnosed with early-stage cervical cancer (FIGO stages IB1-IIA1, excluding FIGO IB3) with negative sentinel lymph node biopsy (SNB) confirmed by ultrastaging.

The main questions it aims to answer are:

Is there a difference in overall survival (OS) and progression-free survival (PFS) between laparoscopic and abdominal radical hysterectomy? Are postoperative complication rates and recurrence patterns comparable between the two surgical approaches?

Researchers will compare outcomes in patients undergoing radical laparoscopic hysterectomy versus abdominal hysterectomy to assess differences in survival, complications, and recurrence.

Participants will:

Have undergone radical hysterectomy (type B or C per Querleu-Morrow classification), preceded optionally by conization, with the use of uterine manipulators and absence of vaginal cuff protection explicitly excluded; Have had SNB as part of surgical staging; Be followed every 6 months for 5 years; Undergo clinical gynecologic examination and transvaginal and/or transabdominal ultrasound during follow-up; Undergo additional imaging (CT and/or pelvic MRI) in case of symptoms suggestive of recurrence.

All participants will follow standard post-treatment surveillance. No additional interventions beyond routine follow-up will be performed. Data on OS, PFS, complications (within 30 and 60 days postoperatively, classified by Clavien-Dindo), duration of surgery, recurrence site, and demographic characteristics will be collected.

DETAILED DESCRIPTION:
Scientific Description This is a retrospective observational study with prospective follow-up designed to evaluate the long-term oncologic safety and perioperative outcomes of radical laparoscopic hysterectomy compared to abdominal (open) radical hysterectomy in women with early-stage cervical cancer. The study specifically addresses surgical management practices adopted after the publication of the Laparoscopic Approach to Cervical Cancer (LACC) trial, which reported inferior oncologic outcomes associated with minimally invasive surgery (MIS) for radical hysterectomy.

The primary objective of this study is to compare overall survival (OS) and progression-free survival (PFS) between the two surgical approaches. Secondary objectives include assessment of short-term surgical morbidity, recurrence patterns, and demographic and clinical factors potentially associated with adverse outcomes.

Study Population Eligible participants will be adult (≥18 years), legally competent women diagnosed with early-stage cervical cancer, defined as FIGO 2018 stages IB1 to IIA1, excluding IB3 tumors. All patients must have negative sentinel lymph node biopsy (SNB) results confirmed by ultrastaging.

To ensure homogeneity and minimize confounding associated with surgical technique, strict intraoperative criteria will be applied:

Use of a uterine manipulator is not permitted; A protective vaginal cuff closure maneuver (e.g., by suture, clamp, or stapler) must be performed to prevent tumor spillage during colpotomy; SNB may be performed as a first step, followed by radical hysterectomy classified as type B or C according to the Querleu-Morrow classification; Preoperative conization is allowed but not mandatory.

Study Design This is a retrospective cohort study with prospective follow-up. Surgical and perioperative data will be collected retrospectively from medical records. Eligible patients who underwent radical hysterectomy by either laparoscopic or abdominal approach in the post-LACC era will be identified and included.

Prospective follow-up will be conducted over a minimum period of 5 years, with evaluations scheduled at 6-month intervals.

Each follow-up visit will include:

Gynecological examination and transvaginal and/or transabdominal ultrasound; In symptomatic patients, additional imaging including contrast-enhanced CT scan of the chest, abdomen, and pelvis, and pelvic MRI as clinically indicated.

Endpoints

Primary endpoints:

Overall survival (OS): Time from radical hysterectomy to death from any cause. Progression-free survival (PFS): Time from radical hysterectomy to first documented recurrence or death.

Secondary endpoints:

Surgical complication rates within 30 and 60 days postoperatively, categorized using the Clavien-Dindo classification; Anatomic site and mode of recurrence (local, regional, or distant); Duration of surgery; Demographic and clinical variables, including age, BMI, tumor size, histologic subtype, and lymphovascular space invasion (LVSI).

Data Collection and Management Data will be extracted from patient medical records, surgical reports, pathology reports, and follow-up documentation. No study-specific interventions will be introduced beyond the standard follow-up protocol consistent with national and institutional guidelines for cervical cancer surveillance.

All clinical, surgical, and outcome data will be anonymized and stored securely. Data analysis will involve time-to-event methods (Kaplan-Meier curves, Cox proportional hazards models) and comparative statistics (e.g., chi-square, t-test, or non-parametric equivalents as appropriate).

Scientific Rationale The LACC trial demonstrated inferior disease-free and overall survival outcomes for minimally invasive radical hysterectomy compared to open surgery, which prompted a global shift in surgical practice. However, methodological concerns-including inconsistent use of uterine manipulators, absence of protective colpotomy techniques, and variability in surgeon experience-may have influenced the observed outcomes.

This study seeks to investigate whether meticulous surgical technique, standardized intraoperative precautions (such as omission of uterine manipulators and protective closure of the vaginal cuff), and proper patient selection (i.e., early-stage tumors with negative SNB) can mitigate the risks previously associated with the laparoscopic approach.

By comparing outcomes in a well-defined cohort treated after dissemination of the LACC trial results, this study aims to provide contemporary, real-world data on the oncologic safety of laparoscopic radical hysterectomy in selected early-stage cervical cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Women undergoing radical hysterectomy type B or C according to the Querleu-Morrow classification for early-stage cervical cancer (FIGO stages IB1-IIA1, excluding FIGO IB3 between November 2018 and August 2025 Not using manipulator during surgery Vaginal cuff protective maneuver during surgery Conization before surgery (optional) SNB as a first stage of treatment (optional)

Exclusion Criteria:

Women undergoing surgery for advanced stage cervical cancer (FIGO >IIA1) or FIGO IB3 Metastasis detected in sentinel node biopsy (confirmed in ultrastaging) ECOG>2 Not willing to participate in the study Not willing to undergo CT-scans or gynecological examinations

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants will include adult, legally competent women undergoing surgery for early-stage cervical cancer (FIGO stages IB1-IIA, excluding FIGO IB3) with negative ultrastaging in sentinel node biopsy (SNB). Not using manipulator and vaginal cuff protective maneuver (either by clamping, suture from abdominal or vaginal site or with stapler) are mandatory. SNB might be a first step of the procedure followed by radical hysterectomy type B or C according to the Querleu-Morrow classification. Conization before hysterectomy is optional. Radical hysterectomy is mandatory procedure in inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
OS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Overall survival

SECONDARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Progression-free survival
Complications | From enrollment to the 30 and 60 days postoperatively
  Complication rate based on Clavien-Dindo Classification
Recurrence | Through study completion, an average of 6 months
  site of the recurrence

CONTACTS AND LOCATIONS:
Locations (5):
- Poland (5):
  - Uniwersyteckie Centrum Onkologii, Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - Department of Gynaecology, Obstetrics and Gynaecological Oncology, University Clinical Centre, Medical University of Silesia, Katowice
  - Klinika Ginekologii, Świętokrzyskie Centrum Onkologii, Samodzielny Publiczny Zakład Opieki Zdrowotnej, Kielce
  - Oddział Ginekologii Onkologicznej z Pododdziałem Urologii, Opolskie Centrum Onkologii, Opole
  - Department of Gynaecological Oncology,, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
IPD after anonymizations will be available on request
Supporting Information: Study Protocol
Time Frame: After completion of recruitment
Access Criteria: On request